CLINICAL TRIAL: NCT07000357
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Effect of AZD0780 on Major Adverse Cardiovascular Events in Patients With Established Atherosclerotic Cardiovascular Disease (ASCVD) or at High Risk for a First ASCVD Event
Brief Title: A Phase III Study of AZD0780 on Major Adverse CV Events in Patients With a History of ASCVD Events or at High Risk for a First Event
Acronym: AZURE-Outcomes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7960C00015; 2025-520519-14 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-05-30; First posted 2025-06-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease
Keywords: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: International, multi-centre, randomised, double-blind, placebo-controlled, parallel-group, event-driven
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD0780 (Experimental): Participants will receive oral AZD0780 once daily
  Interventions: Drug: AZD0780
- Placebo (Placebo Comparator): Participants will receive oral placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0780 — Participants will receive oral AZD0780 once daily
  Arms: AZD0780
Drug: Placebo — Participants will receive oral placebo once daily
  Arms: Placebo

SUMMARY:
The purpose of this phase 3, randomized, placebo controlled, event-driven study is to assess the effect of AZD0780, an oral PCSK9 inhibitor, compared with placebo in reducing the risk of MACE-PLUS in patients with established ASCVD or at high risk for a first ASCVD event. The effect of AZD0780 vs placebo on the risk of MACE-PLUS will be evaluated from randomisation until the primary analysis censoring date (PACD). The Study Closure Visit will be scheduled to occur after the PACD and will be the final visit for each participant in the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following:

  1. Participants with history of an ASCVD event: Participants ≥ 18 years of age at the time of signing the ICF with a history of ASCVD defined as ACS ≥ 1 month to ≤ 12 months prior to randomisation, ischaemic stroke suspected to be due to atherosclerotic vascular disease ≥ 1 month to ≤ 12 months prior to randomisation, or revascularisation for symptomatic lower limb PAD any time prior to screening

     Additional risk factors based on the level of the LDL-C:
     * Participants with an LDL-C ≥ 75 mg/dL (≥ 1.9 mmol/L) need to have at least one of the other additional risk factors (i to viii) below.

       i) T2DM requiring ongoing medical therapy ii) Age ≥ 65 years v) Previous above ankle amputation due to PAD vi) Previous diagnosis of non-end stage CKD
  2. Participants at increased risk of a first ASCVD event: Male participant ≥ 50 years of age or female participant ≥ 55 years of age at the time of signing the ICF with LDL-C ≥ 100 mg/dL (≥ 2.6 mmol/L) and diagnostic evidence of at least one of the following disease categories (i, ii, or iii):

  i) Significant atherosclerotic artery disease ii) High-risk Type 1 or Type 2 diabetes mellitus with manifestation of end-organ disease (diabetic nephropathy, retinopathy, neuropathy or an ABI outside the normal range [0.9 to 1.4]) iii) Documented atherosclerosis of less significance

For (ii) and (iii), participants need to have at least one of the additional risk factors below:

1. CKD with eGFR x mL/min/1.73 m2
2. Current tobacco use
3. Age ≥ 65
4. T2DM (if included on the less significant atherosclerosis criterion iii)

   * Participants should receive a background lipid lowering regimen anticipated to achieve at least a ~50% reduction in LDL-C. Except in cases of intolerance, the regimen should include a high intensity statin therapy or lower intensity statin therapy in combination with an oral agent with proven outcome benefit (eg, ezetimibe and/or bempedoic acid).

Participants must achieve a stable background lipid lowering therapy > 28 days before screening.

Exclusion criteria:

* Any underlying known disease, or condition including homozygous familial hypercholesterolaemia, or LDL or plasma apheresis within 12 months prior to randomisation, that, in the opinion of the investigator, might interfere with the interpretation of the clinical study results.
* Any revascularisation procedure planned within the next 3 months.
* Available imaging assessment within the last 3 years showing either coronary calcium score of zero, or a coronary computed tomography angiography with no atherosclerosis.
* Calculated eGFR < 15 mL /min/1.73 m2 at screening.
* Any laboratory values with the following deviations at screening:

  * AST or ALT > 3 × ULN
  * TBL > 2 × ULN (except for participants with Gilbert's syndrome where TBL 3 × ULN is acceptable provided direct bilirubin < 1.5 × ULN)
  * Fasting triglycerides ≥ 400 mg/dL (≥ 4.52 mmol/L).
  * Creatine kinase > 5 × ULN
  * Urine albumin/creatinine ratio ≥ 500 mg/g
* Uncontrolled T2DM defined as HbA1c ≥ 9.5% at screening.
* Inadequately treated hypothyroidism defined as TSH > 1.5 × ULN at screening or participants whose thyroid replacement therapy was initiated or modified within the last 3 months prior to screening.
* Use of mipomersen or lomitapide (cholesterol-lowering medications) within 12 months of screening or planned use during the study.
* Use of gemfibrozil within one week prior to the Screening Visit or planned use during the study.
* Use of PCSK9 inhibitors: evolocumab/alirocumab within 12 weeks of the Screening Visit or planned use during the study, or inclisiran within 18 months of the Screening Visit or planned use during the study, or any other approved PCSK9 inhibitor use within 5 half lives prior to the Screening Visit or planned use during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15100 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2029-10-26 (Estimated); Study Completion 2029-10-26 (Estimated)

PRIMARY OUTCOMES:
Time to first event of any component of MACE-PLUS | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of MACE-PLUS (the composite of CV death, myocardial infarction [MI], ischaemic stroke, acute lower limb ischaemia, major amputation of a vascular aetiology, and urgent arterial revascularisation)

SECONDARY OUTCOMES:
Time to first event of any component of 3P MACE | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of 3-point (3P)-MACE (the composite of CV death, MI, and ischaemic stroke)
Time to first event of any component of MACE PLUS | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of MACE-PLUS in patients with a history of ASCVD
Time to first event of MI | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of MI
Time to first event of urgent coronary revascularisation | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of urgent coronary revascularisation
Time to CV death | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of CV death
Time to first event of MALE | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of major adverse limb event (MALE) (the composite of acute lower limb ischaemia, major amputation of vascular aetiology, and urgent lower extremity revascularisation)
Time to all-cause mortality | Up to approximately 54 months
  To compare the effect of treatment with AZD0780 to placebo in reducing the risk of all-cause mortality

CONTACTS AND LOCATIONS:
Locations (876):
- United States (237):
  - Research Site, Birmingham, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Saraland, Alabama
  - Research Site, Vestavia Hills, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Canoga Park, California
  - Research Site, Castroville, California
  - Research Site, Chula Vista, California
  - Research Site, Fountain Valley, California
  - Research Site, Garden Grove, California
  - Research Site, Lake Forest, California
  - Research Site, Lancaster, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Monterey Park, California
  - Research Site, Newport Beach, California
  - Research Site, Norco, California
  - Research Site, Northridge, California
  - Research Site, Pomona, California
  - Research Site, Poway, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, Santa Ana, California
  - Research Site, Tarzana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, West Hills, California
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Crystal River, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake City, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Largo, Florida
  - Research Site, Longwood, Florida
  - Research Site, Maitland, Florida
  - Research Site, Margate, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Seminole, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Hinesville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Peachtree Corners, Georgia
  - Research Site, Riverdale, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Union City, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Tinley Park, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Carmel, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Versailles, Kentucky
  - Research Site, Bossier City, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Hammond, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Lanham, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Pikesville, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Brookline, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Dearborn Heights, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Hazelwood, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Elkhorn, Nebraska
  - Research Site, Fremont, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Laurelton, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Lima, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Munroe Falls, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Horsham, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, West Chester, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Fort Mill, South Carolina
  - Research Site, Mauldin, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Elizabethton, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Morristown, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Brownsville, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, El Paso, Texas
  - Research Site, Euless, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Irving, Texas
  - Research Site, Katy, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Paris, Texas
  - Research Site, Pearland, Texas
  - Research Site, Pharr, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Temple, Texas
  - Research Site, Tomball, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Bountiful, Utah
  - Research Site, Ogden, Utah
  - Research Site, Roy, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, White River Junction, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Hopewell, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Redmond, Washington
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (15):
  - Research Site, CABA
  - Research Site, Ciudad Autonoma de Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Ciudad de Rosario
  - Research Site, Córdoba
  - Research Site, Godoy Cruz
  - Research Site, Lanús Este
  - Research Site, Mar del Plata
  - Research Site, Nueva Córdoba
  - Research Site, Rosario
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Rosa
  - Research Site, Zárate
- Brazil (26):
  - Research Site, Aracaju
  - Research Site, Barretos
  - Research Site, Belém
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Criciúma
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Juiz de Fora
  - Research Site, Marília
  - Research Site, Natal
  - Research Site, Ponta Grossa
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, São Caetano do Sul
  - Research Site, São José do Rio Preto
  - Research Site, São José dos Campos
  - Research Site, São Paulo
  - Research Site, Tatuí
  - Research Site, Teresina
  - Research Site, Uberlândia
  - Research Site, Vila Velha
- Bulgaria (7):
  - Research Site, Botevgrad
  - Research Site, Haskovo
  - Research Site, Pernik
  - Research Site, Plovdiv
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (23):
  - Research Site, Red Deer, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (11):
  - Research Site, Antofagasta
  - Research Site, Chillán
  - Research Site, Concepción
  - Research Site, Independencia
  - Research Site, Las Condes
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Valdivia
  - Research Site, Victoria
  - Research Site, Viña del Mar
- China (62):
  - Research Site, Anyang
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Daqing
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Ha’erbin
  - Research Site, Hefei
  - Research Site, Heze
  - Research Site, Hohhot
  - Research Site, Huaian
  - Research Site, Huangshi
  - Research Site, Huizhou
  - Research Site, Jiangmen
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Jinzhou Shi
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Lishui
  - Research Site, Liuchow
  - Research Site, Luoyang
  - Research Site, Meihekou
  - Research Site, Meizhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Neijiang
  - Research Site, Pinggu
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shaoguan Shi
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Siping
  - Research Site, Suining
  - Research Site, Suzhou
  - Research Site, Taian
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wanzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xianyang
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yueyang
  - Research Site, Yuncheng
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
  - Research Site, Zhenjiang
  - Research Site, Zhuhai
  - Research Site, Zhuozhou
  - Research Site, Zibo
- Colombia (9):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Cartagena
  - Research Site, Chía
  - Research Site, Ibagué
  - Research Site, Medellín
  - Research Site, Pasto
- Czechia (16):
  - Research Site, Benátky nad Jizerou
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, Broumov
  - Research Site, Bruntál
  - Research Site, Česká Třebová
  - Research Site, České Budějovice
  - Research Site, Český Krumlov
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Ostrava-Dubina
  - Research Site, Prague
  - Research Site, Pribram VIII
  - Research Site, Svitavy
  - Research Site, Třebíč
  - Research Site, Zlín
- Denmark (13):
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Gandrup
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, Roskilde
  - Research Site, Slagelse
  - Research Site, Svendborg
  - Research Site, Vejle
  - Research Site, Viborg
- France (20):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Narbonne
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valenciennes
- Germany (70):
  - Research Site, Amberg
  - Research Site, Bad Friedrichshall
  - Research Site, Bad Homburg
  - Research Site, Bad Oeynhausen
  - Research Site, Bechhofen
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bonn
  - Research Site, Brandenburg
  - Research Site, Bremen
  - Research Site, Bruchsal
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Fulda
  - Research Site, Göttingen
  - Research Site, Greifswald
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Haßloch
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Herne
  - Research Site, Hohenmölsen
  - Research Site, Jena
  - Research Site, Jerichow
  - Research Site, Kaiserslautern
  - Research Site, Kamp-Lintfort
  - Research Site, Karlsbad
  - Research Site, Karlsruhe
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Lichtenberg
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mainz A. Rhein
  - Research Site, Mannheim
  - Research Site, Markkleeberg
  - Research Site, Munich
  - Research Site, Mühldorf A. Inn
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Obertshausen
  - Research Site, Offenbach
  - Research Site, Oranienburg
  - Research Site, Osnabrück
  - Research Site, Papenburg
  - Research Site, Potsdam
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Rotenburg A.d. Fulda
  - Research Site, Rüsselsheim am Main
  - Research Site, Schwerin
  - Research Site, Speyer
  - Research Site, Stuhr
  - Research Site, Stuttgart
  - Research Site, Trier
  - Research Site, Villingen-Schwenningen
  - Research Site, Weinheim
  - Research Site, Wermsdorf
  - Research Site, Wiesbaden
  - Research Site, Witten
- Greece (8):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Chios
  - Research Site, Heraklion
  - Research Site, Heraklio
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (16):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Encs
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Nyíregyháza-Sóstóhegy
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- India (20):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Dwārka
  - Research Site, Gūrgaon
  - Research Site, Hydarabad
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Ludhiana
  - Research Site, Manipal
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, New Dehli
  - Research Site, New Delhi
  - Research Site, Vadodara
  - Research Site, Vijayawada
- Italy (24):
  - Research Site, Altamura
  - Research Site, Arzignano
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Caserta
  - Research Site, Catania
  - Research Site, Cona
  - Research Site, Foggia
  - Research Site, Genoa
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pordenone
  - Research Site, Rimini
  - Research Site, Rivoli
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Salerno
  - Research Site, Torino
- Japan (60):
  - Research Site, Ami-machi
  - Research Site, Asahi-shi
  - Research Site, Asahikawa-shi
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Fukui-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiyamato-shi
  - Research Site, Hiroshima
  - Research Site, Ichikawa-shi
  - Research Site, Kakegawa-shi
  - Research Site, Kamakura
  - Research Site, Kanazawa
  - Research Site, Kanoya-shi
  - Research Site, Kashihara-shi
  - Research Site, Kashiwara-shi
  - Research Site, Kasuga-shi
  - Research Site, Kasuya-gun
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyushu
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Komatsu-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Machida-shi
  - Research Site, Matsuyama
  - Research Site, Minatoku
  - Research Site, Minokamo Shi
  - Research Site, Miyakonojo-shi
  - Research Site, Miyazaki
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Nakagami-gun
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Osaka
  - Research Site, Ōbu
  - Research Site, Ōita
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Suita-shi
  - Research Site, Suwa-shi
  - Research Site, Tamanashi
  - Research Site, Tanabe-shi
  - Research Site, Tokushima
  - Research Site, Toride-shi
  - Research Site, Toyama
  - Research Site, Toyota
  - Research Site, Tsu
  - Research Site, Tsukuba
  - Research Site, Urasoe-Shi
  - Research Site, Urayasu-shi
  - Research Site, Ushiku-shi
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- Malaysia (13):
  - Research Site, Alor Star
  - Research Site, Cheras
  - Research Site, George Town
  - Research Site, Kajang
  - Research Site, Kota Kinabalu
  - Research Site, Kota Samarahan
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Kubang Kerian
  - Research Site, Kuching
  - Research Site, Sarawak Miri
  - Research Site, Seri Manjung
- Mexico (15):
  - Research Site, Acapulco
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Querétaro
  - Research Site, San Juan del Río
  - Research Site, Torreón
  - Research Site, Veracruz
  - Research Site, Zapopan
- New Zealand (13):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Ebdentown
  - Research Site, Grafton
  - Research Site, Hamilton
  - Research Site, Hastings
  - Research Site, Hutt Central
  - Research Site, New Lynn
  - Research Site, Palmerston North Central
  - Research Site, Papatoetoe
  - Research Site, Pukekohe
  - Research Site, Rotorua
  - Research Site, Woodhill
- Peru (7):
  - Research Site, Bellavista
  - Research Site, Chorrillos
  - Research Site, Lima
  - Research Site, Miraflores
  - Research Site, Piura
  - Research Site, San Isidro
  - Research Site, Wanchac
- Philippines (14):
  - Research Site, Angeles City
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Dasmariñas
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Laguna
  - Research Site, Manadaluyong City
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, San Juan City
  - Research Site, Tacloban City
- Poland (20):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Jelenia Góra
  - Research Site, Katowice
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrów Mazowiecka
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Puerto Rico (2):
  - Research Site, Mayagüez
  - Research Site, San Juan
- Romania (9):
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Satu Mare
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Slovakia (13):
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Malacky
  - Research Site, Nitra
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Šamorín
  - Research Site, Trnava
  - Research Site, Vinica
  - Research Site, Žilina
- South Africa (19):
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Brackenfell
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Kimberley
  - Research Site, Middelbrug
  - Research Site, Midrand
  - Research Site, Paarl
  - Research Site, Panorama
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Tygervalley
  - Research Site, Umhlanga
  - Research Site, Wentworth
- South Korea (12):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Changwon-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Gwangmyeong
  - Research Site, Junggu
  - Research Site, Seoul
  - Research Site, Suncheon
  - Research Site, Yongin-si
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Sanlúcar de Barrameda (Cádiz)
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Villamartín (Cádiz)
- Sweden (9):
  - Research Site, Alingsås
  - Research Site, Falun
  - Research Site, Huddinge
  - Research Site, Lund
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Västerås
- Taiwan (10):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yilan
- Thailand (9):
  - Research Site, Bangkok
  - Research Site, Banphaeo
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Klong Luang
  - Research Site, Mueang
  - Research Site, Nakhon Ratchasima
  - Research Site, Udon Thani
- Turkey (Türkiye) (14):
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Çanakkale
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Kazımkarabekir
  - Research Site, Kütahya
  - Research Site, Muğla
  - Research Site, Odunpazari
  - Research Site, Tokat Province
  - Research Site, Yenimahalle
- Ukraine (7):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (30):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Bridgend
  - Research Site, Bristol
  - Research Site, Calow
  - Research Site, Cambridge
  - Research Site, Chippenham
  - Research Site, Congleton
  - Research Site, Dudley
  - Research Site, Dundee
  - Research Site, Enfield
  - Research Site, Gateshead
  - Research Site, Glasgow
  - Research Site, Harefield
  - Research Site, Isleworth
  - Research Site, Kings Lynn
  - Research Site, Lincoln
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Middlesbrough
  - Research Site, Middlesex
  - Research Site, Milton Keynes
  - Research Site, Newcastle upon Tyne
  - Research Site, Poole
  - Research Site, Portsmouth
  - Research Site, Sheffield
  - Research Site, Wakefield
  - Research Site, Worcester
  - Research Site, Wrexham
  - Research Site, Yeovil
- Vietnam (9):
  - Research Site, Can Tho
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Hồ Chí Minh
  - Research Site, Huế
  - Research Site, Vĩnh Yên

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/